CLINICAL TRIAL: NCT05806528
Title: Role of Placental Invasion Index in Decision Making of Placenta Accreta
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mariam Sabry Mahmoud, Resident at GYN/OBS department, Sohag University
Other Study IDs: Soh-Med-23-03-03MS
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ultrasound — Use ultrasound to make placental invasion index

SUMMARY:
This study will be conducted on women who have a diagnosis of placenta previ and using ultrasound to make the placenta invasion index and compare the accuracy of the diagnosis during the caesarean section whether it is accreta or not with determining the site and depth of invasion

DETAILED DESCRIPTION:
This study will be conducted on women who have a diagnosis of placenta previ and using ultrasound to make the placenta invasion index and compare the accuracy of the diagnosis during the caesarean section whether it is accreta or not with determining the site and depth of invasion and whether there is injury occurred in the urinary system and Determining the amount of blood transfusion and admission of intensive care, or whether the patient death

ELIGIBILITY:
Inclusion Criteria:

* all placenta previa and low laying placenta will be included

Exclusion Criteria:

* patient with sever attack

Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant female
Study Population: Pregnant female with placenta previa
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Role of placental invasion index in decision making of placenta accreta | 1 year
  Use of ultrasound to make placenta invasion index and compare it intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Mariam S Mahmoud, Resident, Principal Investigator — Sohag univesity hospital

IPD SHARING:
Plan to Share IPD: Undecided